CLINICAL TRIAL: NCT05543122
Title: Drugs in Breast Milk
Brief Title: Drug Concentrations in Breast Milk and Prediction of Blood Levels of the Breastfed Infants
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: St. Justine's Hospital (Other); University of Waterloo (Other)
Responsible Party: Principal Investigator, Shinya Ito, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000062184
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding | interventions — Bupropion; brivaracetam; Escitalopram; Fluconazole; Lacosamide; Lamotrigine; Levetiracetam; Methotrexate; Ezetimibe; Dexetimide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — breast milk samples, optional DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breastfeeding women: Either of the following drugs at steady state (Atenolol, Bupropion, Brivaracetam, Escitalopram, Fluconazole, Lacosamide, Lamotrigine, Levetiracetam, Methotrexate or Ezetimibe).
  Interventions: Drug: either of Atenolol, Bupropion, Brivaracetam, Escitalopram, Fluconazole, Lacosamide, Lamotrigine, Levetiracetam, Methotrexate or Ezetimibe

INTERVENTIONS:
Drug: either of Atenolol, Bupropion, Brivaracetam, Escitalopram, Fluconazole, Lacosamide, Lamotrigine, Levetiracetam, Methotrexate or Ezetimibe — This is a cohort study of pharmacokinetics of drugs in milk. Participants in the group are those breastfeeding women on the listed drugs at steady state, who are prescribed these drugs for clinical reasons outside this study framework.
  Other Names: Typical brand names include, but not limited to: Tenoretic, Wellbutrin, Zyban, Briviact, Cipralex, Lexapro, Diflucan, Vimpat, Lamictal, Keppra, Trexall, Xatmep, Ezetrol, Nexlizet

SUMMARY:
There is a significant lack of information on drug secretion into milk and infant exposure. As a first step to address this issue, the investigators examine milk concentrations of selected drugs prescribed to breastfeeding women, which lack milk excretion data. Milk data will be analyzed using population pharmacokinetic approaches, when possible, and acquired data of drug concentration profiles in milk will be combined with infant physiologically-based pharmacokinetic (PBPK) models to predict infant exposure levels.

DETAILED DESCRIPTION:
In this study the investigators measure drug concentrations in breast milk (and optional blood) samples collected through sparse and flexible sampling strategy mitigating intense approaches of conventional PK study. Whenever possible, population PK method is used to characterize milk concentration profiles of the selected drugs. The obtained data is further processed through a PBPK model of infant to predict infant drug exposure levels.

The study also includes an optional pharmacogenetic part. This will allow the investigators to understand how variations in genetic composition plays role in breaking down drugs and how it affects the drug transfer into breast milk.

This study is conducted at three sites: Hospital for Sick Children (leading site), CHU Sainte Justine Hospital, Montreal (Study Lab: for drug measurement), and University of Waterloo (Modelling Core: to create computer model).

ELIGIBILITY:
Inclusion Criteria for breastfeeding women

* Age of 18 years or older
* Lactating women taking at least one of the study target drugs per Standard of Care
* Obtained informed consent
* Ability to communicate in English

Exclusion Criteria for breastfeeding women

* Any concomitant medication
* Known pregnancy during PK sampling

Inclusion criteria for their infant

* Older than 1 week
* Healthy

Exclusion criteria for their infant

* Concomitant medical treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lactating women over the age of 18 who are taking one of the study medications at steady state. Potential participants (breastfeeding women) will be identified by the clinics of collaborators and if interested in participation their verbal consent will be obtained to share their contact information with the study team. Participation of breastfed infants of the mother is optional.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
concentrations of target drugs in breast milk | an average of 1 year
  using assays of drug concentrations validated in human milk as a matrix

CONTACTS AND LOCATIONS:
Locations (1):
- Mehzabin Rahman, Toronto, Ontario, Canada